CLINICAL TRIAL: NCT06175052
Title: A Personalized Nutrition Intervention for Adolescent Depression: A Mixed-Methods Pilot
Brief Title: A Personalized Nutrition Intervention for Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Daphne Korczak, Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TeenDiet_Dep
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: adolescents; diet
MeSH Terms: conditions — Depression | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Nutrition (Experimental): This group will receive the nutrition intervention
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Four nutrition counselling sessions conducted over eight weeks, in conjunction with food items to assist in meal preparation and with weekly educational information messages sent via email.

SUMMARY:
This study is being done to test the feasibility of a personalized nutrition eating plan in adolescents with depression. Evidence suggests that dietary quality may affect an individual's mood. A healthy diet includes vegetables, fruit, nuts, seeds, and olive oil, as well as minimally processed whole grains, legumes, and moderate amounts of lean meat, fish, and dairy.

The investigators will examine the feasibility of a personalized nutrition eating plan for children and youth with depression. Previous research has shown that it helps improve depressive symptoms in adults, but it is not clear if the same is true for children and youth.

DETAILED DESCRIPTION:
The proposed 8-week, mixed-methods, single-arm study aims to examine the feasibility of an adjunctive personalized dietary intervention for adolescents with major depressive disorder. The secondary aims are to determine potential barriers and facilitators of implementation and to improve adherence and uptake.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MDD as determined by semi-structured diagnostic interview
* access to the internet and a computer or smart phone
* presence of a parent who is willing to participate

Exclusion Criteria:

* adherent to a high-quality diet at baseline
* presence of an eating disorder, as determined by semi-structured diagnostic interview
* currently participating in other dietary programs or studies
* actively attempting to increase or decrease body weight;
* presence of a chronic medical condition;
* unstable psychiatric condition (e.g., mania, active suicidal ideation)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Baseline, 9 weeks
  Feasibility of Intervention Measure (FIM). The FIM is a self-reported four-item measure scored using a five-point Likert scale ranging from 'completely disagree' (1) to 'completely agree' (5) with higher scores indicating greater acceptability or feasibility. Higher scores indicate greater feasibility with a maximum score of 20.
Acceptability of the Intervention | Baseline, 9 weeks
  Acceptability of Intervention Measure (AIM). The AIM is a self-reported four-item measure scored using a five-point Likert scale ranging from 'completely disagree' (1) to 'completely agree' (5) with higher scores indicating greater acceptability or feasibility. Higher scores indicate greater acceptability with a maximum score of 20.
Feasibility, Acceptability, and Satisfaction of the Intervention | Baseline, 9 weeks
  Feasibility, Acceptability, and Satisfaction are also assessed using semi-structured qualitative interviews pre- and post-study intervention.

SECONDARY OUTCOMES:
Depression symptoms | Baseline, 5 weeks, 9 weeks
  Depression symptoms are assessed using the Centre for Epidemiological Studies Depression Scale for Children (CES-DC), a validated 20-item self-report measure. Participants rated their symptoms on a four-point Likert scale, with higher scores indicating more severe depression symptoms, and a maximum total score of 60.
Dietary Assessment | Baseline, 5 weeks, 9 weeks
  Adolescents' adherence to the personalized nutrition intervention is assessed using the Mediterranean Diet Quality Index for children and adolescents (KIDMED) questionnaire, a 16-item self- or interviewer-administered measure. Scores range from 0-12. A total score of ≤ 3 indicates poor adherence; a score of 4-7 indicates moderate adherence; a score of ≥8 indicates high adherence.
Nutrition Attitudes and Knowledge questionnaire | Baseline, 9 weeks
  Nutrition attitudes and knowledge are assessed using a Nutrition Attitudes and Knowledge questionnaire, designed to evaluate children's understanding of the 2019 Canada Food Guide (CFG). The questionnaire consists of four five-point Likert scale questions to measure positive attitudes about nutrition with higher scores indicating a stronger belief that healthy eating is important and a maximum score of 20. Additionally, 20 multiple-choice and true/false questions relate to CFG food groups (Drinks, Whole Grain Foods, Vegetables and Fruit, and Protein Foods). Higher scores indicate greater nutrition knowledge and the maximum possible score is also 20.
Parent Food Modelling: | Baseline, 9 weeks
  Parental food modelling is evaluated with 10 items adapted from Cullen's scale, each rated on a four-point Likert scale from 'Never' (0) to 'Always' (3) which has been used to predict diet outcomes in adolescent samples. Higher scores signify greater healthful parental food modeling, with a maximum score of 30.
Satisfaction with menu planning | Baseline, 9 weeks
  Satisfaction with menu planning is evaluated through a single item, independently assessed by parents and adolescents using a five-point Likert scale that ranges from 'very dissatisfied' (1) to 'very satisfied' (5).
Satisfaction with nutrition counselling sessions | Baseline, 9 weeks
  Satisfaction with nutrition counseling sessions is evaluated through a single item, independently assessed by parents and adolescents using a five-point Likert scale that ranges from 'very dissatisfied' (1) to 'very satisfied' (5).

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No